CLINICAL TRIAL: NCT03493282
Title: A Pilot Synaptic Vesicle Glycoprotein 2A (SV2A) PET Study to Evaluate the Effect of CT1812 Treatment on Synaptic Density in Participants With Mild to Moderate Alzheimer's Disease
Brief Title: Effect of CT1812 Treatment on Brain Synaptic Density
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cognition Therapeutics (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COG0105; RF1AG057553 (NIH)
Record Dates: First submitted 2018-02-14; First posted 2018-04-10 (Actual); Results first posted 2023-03-01 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 300 mg (Active Comparator): High Dose CT1812
  Interventions: Drug: Active Treatment- CT1812 300 mg
- 100 mg (Active Comparator): Low Dose CT1812
  Interventions: Drug: Active Treatment- CT1812 100 mg
- Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Active Treatment- CT1812 100 mg — CT1812
  Arms: 100 mg
Drug: Active Treatment- CT1812 300 mg — CT1812
  Arms: 300 mg
Drug: Placebo — Matching Placebo
  Arms: Placebo

SUMMARY:
Study to Evaluate the Safety and Tolerability of Oral CT1812 in Subjects with Mild to Moderate Alzheimer's Disease.

DETAILED DESCRIPTION:
This is a single-center, randomized, double-blind, placebo-controlled, parallel group study of two doses of CT1812 in adults with mild to moderate Alzheimer's Disease to evaluate the safety and tolerability of oral CT1812, administered for up 180 days for the Primary study and another 180 days for the double-blind extension study.

Each participant and caregiver participated in a screening period of up to 60 days, followed by the primary double-blind treatment period of 24 weeks (169 days +/-2) followed by an optional double-blind extension treatment period of another 24 weeks (337 days +/-2).

ELIGIBILITY:
Inclusion Criteria:

* Participants may be included in the study only if they meet all of the following criteria:

  1. Men, and women of non-childbearing potential, 50-85 years of age inclusively, with a diagnosis of mild to moderate Alzheimer's disease according to the 2011 NIA-AA criteria and at least a 6 month decline in cognitive function documented in the medical record.

     1. Non-childbearing potential for women is defined as postmenopausal [last natural menses greater than 24 months; in women under age 55, menopausal status will be documented with serum follicle stimulating hormone (FSH) test] or undergone a documented bilateral tubal ligation or hysterectomy.
     2. Male participants who are sexually active with a woman of child-bearing potential must agree to use condoms during the trial and for 3 months after last dose unless the woman is using an acceptable means of birth control. Acceptable forms of birth control include abstinence, birth control pills, or any double combination of: intrauterine device (IUD), male or female condom, diaphragm, sponge, and cervical cap.
  2. Neuroimaging (MRI) obtained during screening consistent with the clinical diagnosis of Alzheimer's disease and without findings of significant exclusionary abnormalities (see exclusion criteria, number 3).
  3. MMSE 18-26 inclusive
  4. A positive amyloid (Pittsburgh imaging compound B) scan at screening, or history of a positive amyloid scan prior to study entry, or prior lumbar puncture with a CSF Abeta concentration consistent with Alzheimer's disease.
  5. Formal education of eight or more years.
  6. Must have a caregiver who sees them at least 10 hours per week, oversees the administration of study drug, and is willing and able to oversee administration of study medication and participate in all clinic visits and some study assessments. The caregiver must provide written informed consent to participate in the study.
  7. Living at home or in the community (assisted living acceptable)
  8. Able to swallow CT1812 capsules.
  9. Stable pharmacological treatment of any other chronic conditions for at least 30 days prior to screening.
  10. Capable of providing either written informed consent or oral assent to the study procedures and for use of protected health information [Health Insurance Portability and Accountability Act (HIPAA) Authorization, if applicable]. If the Participant can provide only assent, their legally authorized representative also must provide written informed consent. Written informed consent also shall be obtained from the responsible caregiver. All consent processes must be undertaken in the presence of a witness and prior to any study procedures.
  11. Must consent to apolipoprotein E (ApoE) genotyping.
  12. Generally healthy with mobility (ambulatory or ambulatory-aided, i.e., walker or cane), vision and hearing (hearing aid permissible) sufficient for compliance with testing procedures.
  13. Able to complete all screening evaluations.

Exclusion Criteria:

* Participants will be excluded from the study if any of the following conditions apply:

  1. Hospitalization or change of chronic concomitant medication within one month prior to screening.
  2. Patients living in a continuous care nursing facility
  3. Screening MRI of the brain indicative of significant abnormality, including, but not limited to, prior hemorrhage or infarct > 1 cm3, >3 lacunar infarcts, cerebral contusion, encephalomalacia, aneurysm, vascular malformation, subdural hematoma, hydrocephalus, space-occupying lesion (e.g. abscess or brain tumor such as meningioma).
  4. MRI incompatible implants and other contraindications for MRI, such as pacemaker, artificial joints, non-removable body piercings, etc. Additionally, participants who meet the following imaging exclusion criteria will not be included in this study:

     1. Claustrophobia that will result in significant anxiety and difficulty lying still for brain imaging (MRI or PET).
     2. Participation in other research studies involving ionizing radiation within one year of the PET scans that would cause the participant to exceed the yearly dose limits for healthy volunteers.
     3. History of IV drug use that would prevent venous access for PET tracer injection.
     4. Severe motor problems that prevent the participant from lying still for brain imaging.
     5. Severe chronic pain (e.g., as the result of rheumatoid arthritis) that would prevent them from lying still during brain imaging.
  5. Clinical or laboratory findings consistent with:

     1. Other primary degenerative dementia, (dementia with Lewy bodies, fronto-temporal dementia, Huntington's disease, Jacob-Creutzfeld Disease, Down's syndrome, etc.)
     2. Other neurodegenerative condition (Parkinson's disease, amyotrophic lateral sclerosis, etc.)
     3. Seizure disorder
     4. Other infectious, metabolic or systemic diseases affecting the central nervous system (syphilis, present hypothyroidism, present vitamin B12 or folate deficiency, other laboratory values) etc.)
  6. A current DSM-V diagnosis of active major depression, schizophrenia or bipolar disorder. Patients with depressive symptoms successfully managed by a stable dose of an antidepressant are allowed entry.
  7. Clinically significant, advanced or unstable disease that may interfere with outcome evaluations, such as:

     1. Chronic liver disease, liver function test abnormalities or other signs of hepatic insufficiency (ALT, AST, total bilirubin > 1.5 x ULN)
     2. Respiratory insufficiency
     3. Renal insufficiency eGFR < 45 mL/min based on the CKD-EPI formula (https://www.questdiagnostics.com/home/physicians/egfr-calculator)Heart disease (myocardial infarction, unstable angina, heart failure, cardiomyopathy within six months before screening)
     4. Bradycardia (<45/min.) or tachycardia (>100/min.)
     5. Poorly managed hypertension (systolic >160 mm Hg and/or diastolic >95 mm Hg) or hypotension (systolic <90 mm Hg and/or diastolic <60 mm Hg)
     6. Uncontrolled diabetes defined by HbA1c >8
  8. History of cancer within 3 years of screening with the exception of fully excised non-melanoma skin cancers or non-metastatic prostate cancer that has been stable for at least 6 months.
  9. Seropositive for human immunodeficiency virus (HIV).
  10. History of acute/chronic hepatitis B or C and/or carriers of hepatitis B (seropositive for Hepatitis B surface antigen [HbsAg] or anti-Hepatitis C [HCV] antibody).
  11. Clinically significant abnormalities in screening laboratory tests, including:

      1. hematocrit less than 33% for males and less than 30% for females
      2. absolute neutrophil cell count of 1200/uL (with the exception of a documented history of a chronic benign neutropenia), or platelet cell count of < 120,000/uL
      3. INR >1.4 or other coagulopathy, confirmed by repeat.
  12. Disability that may prevent the patient from completing all study requirements (e.g. blindness, deafness, severe language difficulty, etc.)
  13. Women who are fertile and of childbearing potential.
  14. Within 4 weeks of screening visit or during the course of the study, concurrent treatment with antipsychotic agents (except risperidone ≤1.5 mg/day, quetiapine ≤100 mg/day, olanzapine ≤5 mg/day, and aripiprazole ≤10 mg/day), antiepileptics (except gabapentin and pregabalin for nonseizure indications), centrally active anti-hypertensive drugs (e.g., clonidine, l-methyl dopa, guanidine, guanfacine, etc.), opiate analgesics, systemic corticosteroids, psychostimulants, antiparkinsonian medications (except for non-parkinsonian indications) and mood stabilizers (e.g., valproate, lithium), sedatives and anxiolytics with the exception that use of short- to medium-acting benzodiazepines for treatment of insomnia is permitted, however, use of sedatives or hypnotics should be avoided for 8 hours before administration of cognitive tests.
  15. Any disorder that could interfere with the absorption, distribution, metabolism or excretion of drugs (e.g. small bowel disease, Crohn's disease, celiac disease, or liver disease.)
  16. Nootropic drugs except stable AD meds (acetylcholinesterase inhibitors and memantine
  17. Suspected or known drug or alcohol abuse, i.e. more than approximately 60 g alcohol (approximately 1 liter of beer or 0.5 liter of wine) per day indicated by elevated MCV significantly above normal value at screening.
  18. Suspected or known allergy to any components of the study treatments.
  19. Enrollment in another investigational study or intake of investigational drug within the previous 30 days or five half-lives of the investigational drug, whichever is longer.
  20. Previous exposure to anti Aβ vaccines
  21. Exposure to passive immunotherapies for AD (e.g. monoclonal antibodies) or BACE inhibitors within the previous 180 days.
  22. Contraindication to undergoing an LP including, but not limited to: inability to tolerate an appropriately flexed position for the time necessary to perform an LP; international normalized ratio (INR) > 1.4 or other coagulopathy; platelet count of < 120,000/μL; infection at the desired lumbar puncture site; taking anti-coagulant medication within 90 days of screening (Note: low dose aspirin is permitted); degenerative arthritis of the lumbar spine; suspected non-communicating hydrocephalus or intracranial mass; prior history of spinal mass or trauma.
  23. Use of NSAIDs more than 2 days in within any 7-day period. Each incidence of use must be recorded in the source and CRF.
  24. Any condition, which in the opinion of the investigator or the sponsor makes the patient unsuitable for inclusion.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2020-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher van Dyck, MD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Dyck CH, Mecca AP, O'Dell RS, Bartlett HH, Diepenbrock NG, Huang Y, Hamby ME, Grundman M, Catalano SM, Caggiano AO, Carson RE. A pilot study to evaluate the effect of CT1812 treatment on synaptic density and other biomarkers in Alzheimer's disease. Alzheimers Res Ther. 2024 Jan 25;16(1):20. doi: 10.1186/s13195-024-01382-2. PMID 38273408

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Location Type: Medical Clinic
Pre-assignment Details: Each participant was screened between Day -60 and Day -1 prior to study drug administration. Participants could choose to participate in the optional double-blind extension treatment period of an additional 24 weeks (337 days +/-2).as well as a follow up visit at 2 weeks after the final treatment visit.
  In the study, 43 patients were enrolled. 23 participants were randomized, and 20 were screen failures.
Groups:
- 300 mg: High Dose CT1812
  Active Treatment- CT1812 300 mg: CT1812 Administered as an oral capsule at dose levels of 300 mg
- 100 mg: Low Dose CT1812
  Active Treatment -CT1812 100 mg: CT1812 Administered as an oral capsule at dose levels of 100 mg
Period: Primary Double-blind Study (180 Days)
Arm/Group | 300 mg | 100 mg | Placebo
Started | 8 | 8 | 7
Completed | 5 | 6 | 6
Not Completed | 3 | 2 | 1
Not completed — Adverse Event | 2 | 2 | 1
Not completed — Subject Moved | 1 | 0 | 0
Period: Double-blind Extension Study (180 Days)
Arm/Group | 300 mg | 100 mg | Placebo
Started | 3 | 6 | 4
Completed | 3 | 6 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 300 mg | 100 mg | Placebo | Total
Number analyzed (Participants) | 8 | 8 | 7 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (10.9) | 68.0 (9.3) | 72.6 (5.8) | 70.0 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 3 | 11
  Male | 4 | 4 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 8 | 7 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 8 | 8 | 6 | 22
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 76.2 (16.9) | 85.6 (5.0) | 74.8 (9.2) | 79.0 (12.1)
Height [Mean (Standard Deviation); unit: cm] | 170.3 (9.9) | 171.4 (12.5) | 172.1 (12.1) | 171.2 (11.0)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.3 (5.7) | 29.5 (4.1) | 25.2 (1.8) | 27.1 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of TEAEs, Related TEAEs, SAEs, and Related SAEs
Description: Number of subjects reported with AEs and the number of AEs reported following administration of the IP summarized by treatment and grouped according to system organ class and preferred term, using descriptive statistics. Summaries of AEs were also presented by severity and by relationship to investigational product. In these summaries, subjects were counted only once per MedDRA term, for the AE of highest severity or least favorable relationship. Summaries were also presented of SAEs and of AEs leading to study withdrawal.
Time Frame: Up to 12 months
Population: Number of Subjects with Treatment Emergent Adverse Events (TEAE)
Measure: Count of Participants; unit: Participants
Groups:
- 300 mg: High Dose CT1812
  CT1812 300 mg
- 100 mg: Low Dose CT1812
  CT1812 100 mg
- All Subjects: Total
Arm/Group | 300 mg | 100 mg | Placebo | All Subjects
Number analyzed (Participants) | 7 | 8 | 6 | 21
Participants
  All TEAEs | 7 | 8 | 6 | 21
  Mild TEAEs | 6 | 4 | 4 | 14
  Moderate TEAEs | 1 | 2 | 1 | 4
  Severe TEAEs | 0 | 2 | 1 | 3
  Related TEAEs | 4 | 3 | 4 | 11
  TEAEs Leading to Treatment Discontinuation | 2 | 2 | 1 | 5
  SAEs | 0 | 3 | 1 | 4
  Related SAEs | 0 | 0 | 0 | 0

2. Secondary Outcome: Change From Baseline in the Imaging of [11C] UCB-J PET Distribution Volume Ratio (DVR)
Description: The Distribution Volume Ratio (DVR) was used to determine the correlations with the cognitive and functional endpoints. For 11C UCB J, the imaging outcome measure was DVR as produced by the Simplified Reference Tissue Model (SRTM2) using dynamic scan data from 0 to 60 min and the whole cerebellum as a reference region. Change from baseline is calculated as the observed value minus the baseline value. A negative change from baseline indicates the progression of disease.
Time Frame: Day 169
Population: All patients who received at least one dose of investigational product and had a post-baseline assessment of any of the cognitive and clinical endpoints.
Measure: Mean (Standard Error); unit: ratio
Groups:
- 100 mg: Low Dose CT1812
  Placebo: Matching Placebo
- Placebo: Matching Placebo
  Active Treatment- CT1812 100 mg: CT1812
Arm/Group | 300 mg | 100 mg | Placebo
Number analyzed (Participants) | 8 | 8 | 7
ratio | -0.043 (0.020) | -0.019 (0.020) | 0.000 (0.020)

3. Secondary Outcome: Change From Baseline in the Imaging of [18F]FDG PET SUV Ratio (SUVR)
Description: For 18F FDG, the primary imaging outcome measure was the SUVR from 60-90 min post injection using whole cerebellum as a reference region. For SUVR, a composite region was determined, including: prefrontal, lateral temporal, posterior cingulate/precuneus, anterior cingulate, lateral parietal, medial temporal, and lateral occipital regions. Change from baseline is calculated as the observed value minus the baseline value. A negative change from baseline indicates the progression of the disease.
Time Frame: Day 169
Population: as for outcome 2
Measure: Mean (Standard Error); unit: ratio
Arm/Group | 300 mg | 100 mg | Placebo
Number analyzed (Participants) | 8 | 8 | 7
ratio | -0.084 (0.017) | -0.044 (0.017) | -0.053 (0.017)

4. Secondary Outcome: Change From Baseline in Volumetric Magnetic Resonance Imaging (MRI)
Description: A composite region of AD affected brain regions was determined, including prefrontal, lateral temporal, posterior cingulate/precuneus, anterior cingulate, lateral parietal, medial temporal, and lateral occipital regions. Baseline is defined as the last measurement taken before the first dose of study drug. Change from baseline is calculated as the observed value minus the baseline value. A negative change from baseline indicates the progression of disease.
Time Frame: Day 169
Population: as for outcome 2
Measure: Mean (Standard Error); unit: cm^3
Arm/Group | 300 mg | 100 mg | Placebo
Number analyzed (Participants) | 8 | 8 | 7
cm^3 | -6.34 (3.49) | -5.59 (3.51) | -13.85 (3.39)

5. Secondary Outcome: Change From Baseline in the Imaging of Functional MRI - Intrinsic Connectivity Contrast (ICC)
Description: For resting state functional MRI, the outcome was ICC. With this approach a map of the total connectivity of each voxel to all other voxels was computed. For ICC, a composite region of AD affected brain regions was determined, including prefrontal, lateral temporal, posterior cingulate/precuneus, anterior cingulate, lateral parietal, medial temporal, and lateral occipital regions. Change from baseline is calculated as the observed value minus the baseline value. A negative change from baseline indicates the progression of disease.
Time Frame: Day 169
Population: as for outcome 2
Measure: Mean (Standard Error); unit: ratio
Arm/Group | 300 mg | 100 mg | Placebo
Number analyzed (Participants) | 8 | 8 | 7
ratio | 0.005 (0.006) | -0.008 (0.006) | -0.006 (0.007)

6. Secondary Outcome: Change From Baseline in the Cerebrospinal Fluid (CSF) Biomarkers
Description: Change from baseline in CSF Aβ 40, CSF Aβ 42, CSF tau, CSF phospho-tau, CSF neurogranin (NRGN), CSF synaptotagmin, CSF(SNAP25), and CSF neurofilament light (NFL). Change from baseline is calculated as the observed value minus the baseline value.
Time Frame: Day 169
Population: The Pharmacodynamic Analysis Set included all subjects who received the investigational product for 6 months and who had both a baseline CSF lumbar puncture and at least one post-dose result for any CSF concentrations.
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | 300 mg | 100 mg | Placebo
Number analyzed (Participants) | 7 | 5 | 6
pg/ml
  Aβ 40 (pg/ml) | -594.0 (381.57) | 517.70 (445.24) | 222.25 (397.27)
  Aβ 42 (pg/ml) | -32.96 (17.55) | 11.62 (21.88) | -13.90 (19.66)
  Tau (pg/ml) | -84.08 (111.96) | 121.22 (131.96) | 36.74 (120.70)
  Phospho-tau (pg/ml) | -7.71 (12.60) | 5.80 (14.91) | -4.67 (13.59)
  NRGN (pg/ml) | -26.79 (16.50) | 14.96 (19.61) | -5.54 (17.77)
  Synaptotagmin (pg/ml) | 0.88 (2.24) | 6.37 (2.64) | 0.68 (2.44)
  SNAP-25 (pg/ml) | -3.15 (1.54) | 0.74 (1.83) | 1.36 (1.66)
  NFL (pg/ml) | 210.77 (149.24) | 265.74 (176.40) | -24.02 (164.56)

7. Secondary Outcome: Change From Baseline ADAS-Cog11 (Alzheimer's Disease Assessment Scale - Cognition Subscale)
Description: The ADAS-Cog11 total score = the sum of all 11 individual items (word recall [10]; commands [5]; constructional praxis [5]; naming objects and fingers [5]; ideational praxis [5]; orientation [8]; word recognition [12]; remembering test instructions [5]; spoken language [5]; word finding [5]; and comprehension of spoken language [5]). The score range for ADAS-cog 11 is 0-70 where a higher score is worse performance. The ADAS-cog methodology is to sum scores for subscales. The results were calculated using the average change from baseline. Baseline is defined as the last measurement taken before the first dose of study drug is administered. Change is calculated as the observed value minus the baseline value. A negative change from baseline indicates improvement.
Time Frame: Day 169
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | 300 mg | 100 mg | Placebo
Number analyzed (Participants) | 8 | 8 | 7
score on a scale | 1.78 (2.101) | 1.28 (2.091) | 1.37 (2.144)

8. Secondary Outcome: Change From Baseline ADAS-Cog13 (Alzheimer's Disease Assessment Scale - Cognition Subscale)
Description: The ADAS-Cog13 total score includes all of the items in the ADAS-Cog11 and the delayed word recall and the number cancellation. For the ADAS-cog 13 the range is 0-85 (score range for Delayed Word Recall [DWR] score is 0-10 and for Number Cancellation [NC] is 0-5, thus the score is ADAS-cog 11[0-70] plus the scores for DWR and NC). A higher score indicates worse performance. The ADAS-cog methodology is to sum scores for subscales. The results were calculated using the average change from baseline. Baseline is defined as the last measurement taken before the first dose of study drug. Change is calculated as the observed value minus the baseline value. A negative change from baseline indicates improvement in cognitive function.
Time Frame: Day 169
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | 300 mg | 100 mg | Placebo
Number analyzed (Participants) | 8 | 8 | 7
score on a scale | 2.62 (2.157) | 1.73 (2.146) | 1.02 (2.178)

9. Secondary Outcome: Change From Baseline ADAS-Cog14 (Alzheimer's Disease Assessment Scale - Cognition Subscale)
Description: The ADAS-Cog14 total score includes all of the items in the ADAS-Cog13 [0-85] and the maze item which has a score range of 0-5. Thus, the total score for the ADAS-cog 14 is 0-90 where again a higher score is worst performance. The ADAS-cog methodology is to sum scores for subscales. The results were calculated using the average change from baseline. Baseline is defined as the last measurement taken before the first dose of study drug is administered. Change is calculated as the observed value minus the baseline value. A negative change from baseline indicates improvement in cognitive function.
Time Frame: Day 169
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | 300 mg | 100 mg | Placebo
Number analyzed (Participants) | 8 | 8 | 7
score on a scale | 1.25 (2.544) | 1.42 (2.245) | 1.65 (2.290)

10. Secondary Outcome: Change From Baseline in ADCS-Activities of Daily Living (ADCS-ADL)
Description: The ADCS-ADL is a 23-item informant-administered assessment of functional impairment in terms of activities of daily living. Informants respond to 23 questions about the subject's involvement and level of performance across items representing daily living. The questions range from basic to instrumental activities of daily living. Each item is rated from the highest level of independent performance to complete loss. The total score range is from 0-78 with lower scores indicating greater functional impairment. A positive change from baseline indicates improvement in function.
  The results were calculated using the average change from baseline. Higher scores mean better outcome.
  Negative mean indicates worsening of function. Positive mean indicates improvement of function.
Time Frame: Day 169
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | 300 mg | 100 mg | Placebo
Number analyzed (Participants) | 8 | 8 | 7
score on a scale | -3.16 (1.646) | -0.31 (1.522) | 2.21 (1.641)

11. Secondary Outcome: Change From Baseline in Mini Mental State Exam (MMSE)
Description: The MMSE assesses several aspects of memory and cognitive functioning including orientation, attention, concentration, comprehension, recall, and praxis. The total possible score is 30, with high scores indicating less impairment. Change from baseline is calculated as the observed value minus the baseline value. A positive change from baseline indicates improvement in cognition.
Time Frame: Day 169
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | 300 mg | 100 mg | Placebo
Number analyzed (Participants) | 8 | 8 | 7
score on a scale | -2.92 (1.540) | -1.26 (1.448) | -0.74 (1.547)

12. Secondary Outcome: Change From Baseline in Clinical Dementia Rating Scale - Sum of Boxes (CDR-SB)
Description: Scores were on a scale of 0 through 3, with 0=no dementia, 0.5=questionable dementia, 1=mild dementia, 2=moderate dementia, and 3=severe dementia. Cognitive and functional abilities that were assessed include Memory; Orientation; Judgment and Problem Solving; Community Affairs; Home and Hobbies; and Personal Care. Memory was considered as the primary driver for scoring and the other categories were secondary. The change from baseline in the CDR-SB total score was analyzed using the mixed model for repeated measures (MMRM). Change from baseline is calculated as the observed value minus the baseline value. Higher scores mean worsening of disease.
Time Frame: Day 169
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | 300 mg | 100 mg | Placebo
Number analyzed (Participants) | 8 | 8 | 7
score on a scale | 0.72 (0.421) | 0.39 (0.399) | 0.17 (0.409)

13. Secondary Outcome: Change From Baseline in Alzheimer's Disease Clinical Study - Clinician Global Impression of Change (ADCS-CGIC)
Description: The scale consists of a format with which a clinician may address clinically relevant overall change, including 15 areas under the domains of cognition, behavior, and social and daily functioning. For ADCS-CGIC, the individual data listing presented the original score on the seven-point scale. In addition, the seven-point score was collapsed to 3 groups, combining scores 1-3 to "Improved", 4 to "No change", and 5-7 to "Worsening". Lower scores indicate improvement.
Time Frame: Day 169
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | 300 mg | 100 mg | Placebo
Number analyzed (Participants) | 8 | 8 | 7
score on a scale | 4.80 (0.279) | 4.50 (0.257) | 4.68 (0.257)

14. Secondary Outcome: Change From Baseline in the Cognitive Composite
Description: The Cognitive composite included:
  1. 6 ADAS-Cog items: word recall, orientation, delayed word recall, word recognition, number cancellation, and maze
  2. 4 Neuropsychological Test Battery (NTB) items: Trail Making Test (TMT) A, Trail Making Test (TMT) B, Category Fluency Test (CFT), Digit span.
  Each individual z-score was calculated by first computing the baseline mean and standard deviation at baseline for all subjects within each individual component. The z-scores were then derived for each subject and timepoint by subtracting the corresponding baseline mean from the observed value and then dividing by the standard deviation at baseline. The sign of the z-score for the following components was reversed when deriving the Composite scores: Word recall, Orientation, Delayed Word Recall, Word Recognition, Maze, TMT A, TMT B.
  Z-score = 0 represents the population at baseline
  Positive Z-score = indicates improvement
  Negative Z-score= indicates worsening
Time Frame: Day169
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Z-Score
Arm/Group | 300 mg | 100 mg | Placebo
Number analyzed (Participants) | 8 | 8 | 7
Z-Score | -0.33 (0.109) | -0.11 (0.102) | -0.10 (0.109)

15. Secondary Outcome: Change From Baseline in the Memory Composite
Description: The memory composite includes 4 ADAS-COG (Alzheimer's Disease Assessment Scale - cognition subscale) items: word recall, orientation, delayed word recall, word recognition. The Memory composite score will be a composite z-score average similar to the Cognitive Composite score but will only be derived using the average of the ADAS-Cog Word Recall, Orientation, Delayed Word Recall, and Word Recognition items. If a subject is missing any of the four items at a timepoint, this composite score will not be derived.
  The score was calculated using z-scores of the items cited above where:
  Z-score = 0 represents the population at baseline.
  Positive Z-score = indicates improvement
  Negative Z-score= indicates worsening
Time Frame: Day169
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Z-score
Arm/Group | 300 mg | 100 mg | Placebo
Number analyzed (Participants) | 8 | 8 | 7
Z-score | -0.49 (0.201) | -0.18 (0.201) | -0.14 (0.198)

16. Secondary Outcome: Change From Baseline in Attention Composite
Description: The Attention composite score included:
  1. 1 ADAS-COG (Alzheimer's Disease Assessment Scale -cognition subscale) item: Number Cancellation
  2. 1 NTB item: Trail Making Test (TMT) A The Attention composite score will be a composite z-score average derived using the average of the Number Cancellation, Maze item from ADAS-Cog 14, and TMT A items. If a subject missed either of the three items at a timepoint, this composite score was derived.
  The score was calculated using z-scores of the items cited above where:
  Z-score = 0 represents the population at baseline.
  Positive Z-score = indicates improvement
  Negative Z-score= indicates worsening
Time Frame: Day 169
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Z-score
Arm/Group | 300 mg | 100 mg | Placebo
Number analyzed (Participants) | 8 | 8 | 7
Z-score | -0.01 (0.158) | 0.15 (0.132) | -0.13 (0.139)

17. Secondary Outcome: Change From Baseline in the Executive Composite
Description: The Executive composite included
  1. 0 ADAS-COG (Alzheimer's Disease Assessment Scale - cognition subscale) items
  2. 3 NTB (Neuropsychological Test Battery) items: CFT (Category Fluency Test), Digit Span, and Trail Making Test (TMT) B The Executive function composite score will be a composite z-score average derived using the average of the CFT Category Fluency Test), Digit Span, and TMT B items. If a subject is missing any of the three items at a timepoint, this composite score will not be derived.
  The score was calculated using z-scores of the items cited above where:
  Z-score = 0 represents the population at baseline.
  Positive Z-score = indicates improvement
  Negative Z-score= indicates worsening
Time Frame: Day 169
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Z-score
Arm/Group | 300 mg | 100 mg | Placebo
Number analyzed (Participants) | 8 | 8 | 7
Z-score | -0.35 (0.366) | 0.66 (0.364) | -0.03 (0.256)

ADVERSE EVENTS:
Time Frame: Up to 12 months
Arm/Group | 300 mg | 100 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 3/8 | 1/7
Other Adverse Events (participants affected / at risk) | 7/8 | 8/8 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 300 mg (N=8) | 100 mg (N=8) | Placebo (N=7)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Thalamic Infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 300 mg (N=8) | 100 mg (N=8) | Placebo (N=7)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral microhaemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (3) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 2 (2) | 2 (2)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Thalamic infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral venous disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 1 (4) | 1 (1)
Carotid endarterectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral Infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ligament Sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Cataract Operation (Surgical and medical procedures) | 0 (0) | 1 (2) | 0 (0)
Gingival graft (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Ureatric Operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-02-03): https://cdn.clinicaltrials.gov/large-docs/82/NCT03493282/Prot_001.pdf
  • Statistical Analysis Plan (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/82/NCT03493282/SAP_002.pdf